CLINICAL TRIAL: NCT03395158
Title: Implementation of New Trauma Triage Criteria and Implications on Under- and Overtriage
Acronym: Traumalert
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: UppsalaUH
Record Dates: First submitted 2017-12-15; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prior alert criteria: Patients who activated full, limited or no alert criteria according to the prior alert criteria
  Interventions: Diagnostic Test: Implementation of new alert criteria
- Present alert criteria: Patients who activated full, limited or no alert criteria according to the present alert criteria
  Interventions: Diagnostic Test: Implementation of new alert criteria

INTERVENTIONS:
Diagnostic Test: Implementation of new alert criteria — The intervention is when the prior alert criteria are replaced by the present alert criteria

SUMMARY:
New trauma alert criteria has been introduced in Sweden, and our aim in this study is to evaluate the outcome of the old and new trauma alert criteria in a cohort of 1.300.000 inhabitants at six hospitals regarding over- and undertriage and number of alerts initiated. The Swedish trauma registry is used to identify eligible patients.

DETAILED DESCRIPTION:
The Swedish trauma registry (SweTrau) was initiated in 2011, and has up to date 40.000 registered patients. In order to evaluate trauma alert criteria implemented during 2017, we plan a prospective stepped wedge trial at six hospitals in the Uppsala/Örebro region. These hospitals register in SweTrau and all had the same alert criteria prior to the implementation of new alert criteria.

A power estimation show the need for 588 patients in each group in order to show a statistical difference between 2-5% undertriage at a 95% CI.

The including hospitals has a population base of 1.300.000 inhabitants, and the annual number of trauma alerts has been about 3.000.

The registry has information about time of trauma, initiated alerts, Injury Severity Score and mechanism of injury suitable for analysis for our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

- All patients registered in SweTrau at all including sites between 1 June 2016 and 1 November 2017

Exclusion Criteria:

* Patients registered due to secondary referral where the initial assessment was performed at another hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients subject to trauma where a trauma alert was initiated OR registered patients subject to trauma without an alert call, but with an Injury Severity Score >15.
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Number of alerts initiated | One year data with intervention
  The total number of trauma alerts initiated in the study group

SECONDARY OUTCOMES:
Analysis of over- and undertriage with the Matrix method | One year data with intervention
  Analyse proportions of patients subject to a full trauma team activation who have an injury severity score <15 (overtriage). Analyse proportion of patients who do not initiate a full trauma team activation but have an injury severity score >15 (undertriage) The Matrix method is a well defined method for analysing resource allocation in trauma triage.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mani, Ass prof, Study Chair — Uppsala University

IPD SHARING:
Plan to Share IPD: No